CLINICAL TRIAL: NCT04295902
Title: Laryngoscopy for Neonatal and Infant aIrway Management wIth Supplemental oxygEn (OPTIMISE): a Multi-center Prospective Randomized Controlled Trial
Brief Title: Laryngoscopy for Neonatal and Infant aIrway Management (Optimise-Trial)
Acronym: Optimise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other); Gaslini Children's Hospital (Other); Children's Hospital of Philadelphia (Other); Montreal Children's Hospital of the MUHC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-02454
Record Dates: First submitted 2020-03-02; First posted 2020-03-05 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Airway Management

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VL-group (Experimental): Tracheal intubation performed with the C-MAC indirect videolaryngoscope (Karl Storz, Germany) with blades Miller nr 0 and Miller nr 1.
  Interventions: Device: C-MAC indirect videolaryngoscope with blades Miller nr 0 and Miller nr 1.
- DL-group (Active Comparator): Tracheal intubation performed with a standard direct laryngoscope, with standard blades Miller nr 0 and Miller nr 1
  Interventions: Device: Direct laryngoscope with blades Miller nr 0 and Miller nr 1.

INTERVENTIONS:
Device: C-MAC indirect videolaryngoscope with blades Miller nr 0 and Miller nr 1. — Tracheal intubation performed with the C-MAC indirect videolaryngoscope (Karl Storz, Tuttlingen, Germany) with blades Miller nr 0 and Miller nr 1.
  Other Names: C-Mac Videolaryngoscope
  Arms: VL-group
Device: Direct laryngoscope with blades Miller nr 0 and Miller nr 1. — Tracheal intubation performed with a standard direct laryngoscope, with standard blades Miller nr 0 and Miller nr 1
  Other Names: Standard direct laryngoscope
  Arms: DL-group

SUMMARY:
The objective of this study is to compare tracheal intubation first attempt success rate with the C-MAC indirect videolaryngoscope (Karl Storz, Germany) using a Miller-Blade nr 0 or nr 1 compared to a standard direct laryngoscope with standard blades Miller nr 0 and Miller nr 1 with oxygen supplementation either in the operating room or intensive care to demonstrate that with oxygen supplementation the difference in the first-attempt success rate in favor of VL is negligible

DETAILED DESCRIPTION:
Eligible children will be prepared for intubation according to the local SOPs of the pediatric anesthesia or pediatric intensive care departments. Mandatory monitoring will consist of: SpO2, HR, NIBP.

Induction of anesthesia: All children included in this protocol will be pre-oxygenated before induction of anesthesia for one minute through face-mask with FiO2 = 1.0 and flow rates of 6-10L/min. The induction of anesthesia for tracheal intubation will be performed using a combination of sedative/hypnotic drugs, opioids and non-depolarizing muscle relaxant.

The following medications will be mandatory as per protocol:

* A non-depolarizing muscle relaxant (NDMR) drug (Rocuronium 0.5-1 mg/kg, Cis-Atracurium 0.2-0.5 mg/kg, Vecuronium 0.1 mg/kg, or succinylcholine 2 mg/kg).
* One or more of the following hypnotic agents (Thiopentone 4-7 mg/kg, Ketamine 0.5-2 mg/kg, Propofol 1-4 mg/kg, Midazolam 0.5-1 mg/kg, Sevoflurane up to 8%).

An opioid drug and anticholinergic can be chosen and administered at the discretion of the anesthetist in charge

Before intubation: After induction of anesthesia and the administration of a muscle relaxant drug, bag-mask ventilation with FiO2 = 1.0 (flow rates of 6-10 Lmin-1) will be performed for 60 seconds until apnea sets in. After induction all patients will be paralysed with e.g. 0.5-1 mg/kg of rocuronium (2 x ED95 (standard intubation dose)) to facilitate airway management. Neuromuscular blockade will be assessed by train-of-four (TOF) monitoring. Thereafter oxygen administration, laryngoscopy and tracheal intubation are performed.

During intubation: The administration of oxygen during intubation is mandatory for every study participant and is standardized as follows:

* Oral intubation: For all orally intubated children, the administration of low-flow oxygen (1 l/kg/min) takes place via conventional neonatal nasal cannula. After administration of low-flow oxygen laryngoscopy and tracheal intubation are performed.
* Nasal intubation: For all nasally intubated children, the administration of low-flow oxygen (1 l/kg/min) takes place direct via nasal tube. The nasal tube is introduced into one of the two nostrils up to the nasopharyngeal space and oxygen is applied to the tube via oxygen cannula. After administration of low-flow oxygen laryngoscopy and tracheal intubation are performed.

For a premature neonate < 1kg an uncuffed tube ID 2.5 will be used. For premature babies and newborn between 1kg and 3.0 kg an uncuffed tube ID 3.0 will be used. For babies > 3.0 kg a cuffed tube ID 3.0 or an uncuffed tube 3.5 will be used. The tube will be either passed through one of the two nostrils and advanced with the help of a Magill-forceps or through the mouth. Based on the group of randomization, the child will be intubated either using the C-MAC videolaryngoscope with a Miller blade 1 (Karl Storz, Germany) or using standard direct laryngoscope, with standard blades Miller nr 0 and Miller nr 1.

Miller blade nr 0 will be used for children < 1 kg. In cases of unexpected difficult intubation, the difficult airway algorithm (14) will be followed. After the first unsuccessful intubation attempt with the randomized device, the investigators encourage to perform a second attempt with the same device but based on the clinical judgment the intubating physician can proceed to an attempt with the same technique, or change the laryngoscope blade size, switch from one technique to another and a maximum of 4 intubation attempts in total will be performed. The last intubation attempt must be performed by the most experienced physician in the room. Additional devices like stylet, bougie, etc, can be used at any stage of the intubation process. If the intubation remains unsuccessful the difficult airway algorithm will be followed and a supraglottic airway device - SAD will be inserted.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients requiring tracheal intubation for elective, semi-elective or urgent surgical and non-surgical indications either in the pediatric operating room, the pediatric or neonatal intensive care unit
* Children aged up to 52 weeks (corrected gestational age), with legal guardians providing written informed consent before the intervention

Exclusion Criteria:

* Prediction of difficult intubation upon physical examination or previous history of difficult intubation, mandating a technique different than direct laryngoscopy to secure the airway
* congenital heart disease mandating FiO2 < 1.0
* cardiopulmonary collapse requiring advanced life support
* intubation for emergency surgical and non-surgical indications

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Tracheal intubation first attempt success rate | 15 minutes
  Primary outcome is tracheal intubation first attempt success rate with the C-MAC indirect videolaryngoscope (Karl Storz, Germany) using a Miller-Blade nr 0 or nr 1 compared to a standard direct laryngoscope with standard blades Miller nr 0 and Miller nr 1.

SECONDARY OUTCOMES:
Occurrence and duration of moderate and severe desaturation | 15 minutes
  Occurrence and duration of moderate and severe desaturation (SpO2 < 90% and SpO2 < 80%), with or without bradycardia, during intubation
Overall number of attempts | 15 minutes
  Overall number of intubation's attempts
Time required for intubation | 5 minutes
  Time required for intubation (in seconds, defined from the first introduction of laryngoscope between the lips till successful lung ventilation defined as positive capnography),
First EtCO2 after successful intubation | 10 minutes
  First EtCO2 after successful intubation
Percentage of Glottic Opening (POGO) score at any attempt of laryngoscopy | 5 minutes
  Percentage of Glottic Opening (POGO) score at any attempt of laryngoscopy
Use of additional devices | 10 minutes
  The need for additional devices used at any step of intubation, the need to switch from one technique to another
Respiratory complications | 24 hours
  Respiratory complications or complications of airway management within the first 24 hours such airway injury, mechanical resuscitation, bleeding, aspiration of gastric contents, post extubation stridor, laryngospasm, bronchospasm, need for High Flow Nasal Oxygen (if not preoperatively on oxygen), need for low flow nasal oxygen (if not preoperatively on oxygen) or need for re-intubation will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Riva, MD, Study Chair — University of Bern
Locations (1):
- University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Riva T, Engelhardt T, Basciani R, Bonfiglio R, Cools E, Fuchs A, Garcia-Marcinkiewicz AG, Greif R, Habre W, Huber M, Petre MA, von Ungern-Sternberg BS, Sommerfield D, Theiler L, Disma N; OPTIMISE Collaboration. Direct versus video laryngoscopy with standard blades for neonatal and infant tracheal intubation with supplemental oxygen: a multicentre, non-inferiority, randomised controlled trial. Lancet Child Adolesc Health. 2023 Feb;7(2):101-111. doi: 10.1016/S2352-4642(22)00313-3. Epub 2022 Nov 24. PMID 36436541